CLINICAL TRIAL: NCT04639128
Title: An Open-Label Randomized Noninferiority Clinical Trial of the Adductor Canal Catheter for Pain Control Post-Total Knee Arthroplasty
Brief Title: Adductor Canal Catheter Effectiveness and Safety Study
Acronym: ACCESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1488728
Record Dates: First submitted 2020-11-05; First posted 2020-11-20 (Actual); Results first posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Total Knee Replacement Surgery
Keywords: analgesia; surgery; device
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- No-Device (No Intervention): No placement of an adductor canal catheter
- Device (Experimental): Placement of an adductor canal catheter
  Interventions: Device: Adductor Canal Catheter

INTERVENTIONS:
Device: Adductor Canal Catheter — The adductor canal catheter is a medical device that consists of a tunneled catheter connected to an analgesic solution-containing reservoir that slowly infuses the anesthetic over the first 2-3 postoperative days
  Arms: Device

SUMMARY:
PRIMARY OBJECTIVE: Compare the effect of usual care with an adductor canal catheter (ACC) containing ropivacaine to the effect of usual care without an ACC on the second-postoperative-day pain levels among patients undergoing elective primary unilateral total knee arthroplasty (TKA)

SECONDARY OBJECTIVES: Among a sample of patients undergoing elective primary unilateral TKA who receive peri-articular anesthetic injections:

1. To compare the overall two-week levels of postoperative pain between those participants randomized to ACCs containing ropivacaine and those participants randomized to usual care without an ACC
2. To compare the use of opioid medications (in mean total morphine milligram equivalents) between those participants randomized to ACCs containing ropivacaine and those participants randomized to usual care without an ACC over the two-week postoperative period
3. To describe the incidence of complications related to ACC placement including infection, displacement, ACC-related clinic or emergency department (ED) visits
4. To conduct exploratory analyses to identify candidate predictors of differential response to the ACC

DETAILED DESCRIPTION:
DESIGN: Randomized, open-label, two-arm, parallel-comparison noninferiority trial

POPULATION: Adults aged >18 years intending to undergo elective primary unilateral TKA at the Kaiser Permanente Northern California (KPNC), San Leandro Medical Center

INTERVENTION: Participants will be randomized to one of two treatment arms:

1. Adductor canal catheter placement in the pre-operative area immediately prior to TKA surgery OR
2. No adductor canal catheter placement

DURATION: The intervention phase will occur between randomization and three days postoperatively (or until the ACC is removed by the participant or the ACC falls out spontaneously among ACC-randomized participants); the primary outcome will be measured on postoperative day 2, secondary pain and medication outcomes will be collected for two weeks postoperatively and the electronic medical record (EMR) will be examined for evidence of adverse events at 30 days postoperatively

SAMPLE SIZE: 118 participants randomized using balanced allocation to the two study arms

ELIGIBILITY:
Inclusion Criteria:

* Intending to undergo elective primary unilateral TKA at the Kaiser Permanente Northern California, San Leandro Medical Center
* Patient ambulates independently

Exclusion Criteria:

* Patient declines use of ACC
* Surgeon decides that an ACC will not be placed for any reason
* Known hypersensitivity to ropivacaine or any alternative anesthetic for ACC use
* Hypersensitivity or inability to tolerate peri-articular injections of clonidine, epinephrine, bupivacaine and ketorolac
* Any evidence of substance-use disorder in past year
* Non-English speaking
* Failure to complete all baseline study instruments prior to surgery
* Requires secondary procedure at time of TKA (e.g., removal of hardware)
* Not intending to use spinal anesthesia for TKA procedure
* Actively enrolled in KPNC chronic-pain program
* Having been prescribed long-acting opioid (e.g., Oxycontin, MS Contin) within 90 days prior to enrollment
* Inability to tolerate any oral NSAID or acetaminophen or any short-acting opioid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2023-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Hinman, MD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente San Leandro, San Leandro, California, United States

IPD SHARING:
Plan to Share IPD: No
Consideration for sharing patient-level data will be made on case-by-case basis via contact with the study PI

REFERENCES:
- [Background] Song MH, Kim BH, Ahn SJ, Yoo SH, Kang SW, Kim YJ, Kim DH. Peri-articular injections of local anaesthesia can replace patient-controlled analgesia after total knee arthroplasty: a randomised controlled study. Int Orthop. 2016 Feb;40(2):295-9. doi: 10.1007/s00264-015-2940-2. Epub 2015 Jul 31. PMID 26227922
- [Background] Manickam B, Perlas A, Duggan E, Brull R, Chan VW, Ramlogan R. Feasibility and efficacy of ultrasound-guided block of the saphenous nerve in the adductor canal. Reg Anesth Pain Med. 2009 Nov-Dec;34(6):578-80. doi: 10.1097/aap.0b013e3181bfbf84. PMID 19916251
- [Background] Kim DH, Lin Y, Goytizolo EA, Kahn RL, Maalouf DB, Manohar A, Patt ML, Goon AK, Lee YY, Ma Y, Yadeau JT. Adductor canal block versus femoral nerve block for total knee arthroplasty: a prospective, randomized, controlled trial. Anesthesiology. 2014 Mar;120(3):540-50. doi: 10.1097/ALN.0000000000000119. PMID 24401769

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | No-Device | Device
Started | 63 | 63
Completed | 60 | 62
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No-Device | Device | Total
Number analyzed (Participants) | 63 | 63 | 126
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (8.6) | 66.5 (9.3) | 66.5 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 35 | 71
  Male | 27 | 28 | 55
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 10 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 11 | 17
  White | 44 | 37 | 81
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 5 | 11
Region of Enrollment [Number; unit: participants]
  United States | 63 | 63 | 126

OUTCOME MEASURES:

1. Primary Outcome: Pain Numerical Rating Scale
Description: Ordinal 0-to-10 point scale of pain severity Minimum value: 0 Maximum value: 10 Higher scores mean more pain
Time Frame: Second postoperative day
Population: Had surgery and able to provide postoperative day-2 pain score
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | No-Device | Device
Number analyzed (Participants) | 60 | 62
score on a scale | 6.38 (0.30) | 5.31 (0.32)

2. Secondary Outcome: Opioid Consumption in the 15-day Postoperative Period
Description: Total number of 5mg oxycodone tablets (provided to all patients on discharge) consumed over the 15-day postoperative period as recorded in the daily pain-and-medication postoperative diary
Time Frame: 15 postoperative days
Population: Numbers of participants do not equal those of the pain-score analyses due to missing data
Measure: Mean (Standard Error); unit: 5mg oxycodone tablets
Arm/Group | No-Device | Device
Number analyzed (Participants) | 47 | 46
5mg oxycodone tablets | 41.9 (4.20) | 46.0 (5.59)

ADVERSE EVENTS:
Time Frame: 30 days postoperatively
Arm/Group | No-Device | Device
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/63
Serious Adverse Events (participants affected / at risk) | 3/63 | 1/63
Other Adverse Events (participants affected / at risk) | 0/63 | 0/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No-Device (N=63) | Device (N=63)
Vertigo (Nervous system disorders) | 0 (0) | 1 (1)
Small-bowel obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Wound dehiscence (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-26): https://cdn.clinicaltrials.gov/large-docs/28/NCT04639128/Prot_SAP_003.pdf
  • Informed Consent Form (2020-10-06): https://cdn.clinicaltrials.gov/large-docs/28/NCT04639128/ICF_001.pdf